CLINICAL TRIAL: NCT03482544
Title: Effect of Orally Pregabalin Given Before Knee Joint Replacement on Reperfusion Injury Which Caused by Bandage
Brief Title: The Effect of Pregabalin Given Preoperatively on the Tourniquet Induced Ischemia-reperfusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Omer Karaca, Assistant Professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA16/10
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Ischemia Reperfusion Injury
Keywords: pregabalin; ischemia reperfusion injury; muscle
MeSH Terms: conditions — Reperfusion Injury | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin Group (Active Comparator): We will give 150 mg pregabalin capsule orally 1 day before surgery and 1 hour before surgery (totally two times) to the pregabalin group patients.
  Interventions: Drug: Pragabalin
- Control Group (Active Comparator): In control group, we will empty the drug material from capsules and give only empty capsules to the control group patients at the same times.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pragabalin — pregabalin 150 mg will be given orally, 1 day and 1 hour before surgery (totally two times), patients in Pregabalin Group.
  Other Names: pregabalin 150 mg, Lyrica, Pfezir, Almanya
  Arms: Pregabalin Group
Other: Placebo — empty capsule will be given orally, 1 day and 1 hour before surgery (totally two times), patients in Control Group.
  Other Names: empty capsule
  Arms: Control Group

SUMMARY:
The application of tourniquet is indispensable for a bloodless surgical area in total knee arthroplasty surgery. The release of tourniquet produces reactive oxygen species which can cause injury and then ischemia-reperfusion injury emerge. Our aim in this study is to investigate effects of pregabalin, GABA analog drug, on the tourniquet induced ischemia-reperfusion injury.

DETAILED DESCRIPTION:
Investigators will randomize patients into two groups. 1) Pregabalin group 2) Control group.

Investigators will give orally pregabalin 150 mg to the pregabalin group patients two times (first dose 1 day before surgery., second dose 1 hour before surgery). On the other hand placebo drug will give to the control group at the same times. Investigators will perform combined spinal epidural anesthesia for surgery and inject 3 cc 0.5% hyperbaric bupivacaine to subarachnoid space. Investigators will take blood samples for measurement of ischemia-reperfusion determinants, immediately before surgery, shortly before tourniquet deflation, and 20 minutes after tourniquet deflation. Then these samples will be analysed by ELISA method.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status I-II
2. Undergoing a total knee arthroplasty surgery
3. Accept neuroaxial anesthesia for surgery

Exclusion Criteria:

1. Any antiepileptic drug use
2. Allergic reaction to pregabalin
3. Severe hepatic, renal or gastrointestinal disorders
4. Psychiatric disorders
5. Pregnant women or breastfeeding
6. NSAID or opioid drug use for a long time
7. Diabetic or other neuropathic pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
ischemia modified albumin | before tournique application,just before tournique release, 20 minutes after tournique release
  changes of ischemia modified albumin
total oxidant status | before tournique application, just before tournique release, 20 minutes after tournique release
  changes of total oxidant status
total antioxidant status | before tournique application, just before tournique release, 20 minutes after tournique release
  changes of total antioxidant status

SECONDARY OUTCOMES:
catalase | before tournique application, just before tournique release, 20 minutes after tournique release
  changes of catalase

CONTACTS AND LOCATIONS:
Overall Officials: Omer Karaca, Assist.Prof, Principal Investigator — Baskent University
Locations (1):
- Baskent University, Konya, Turkey (Türkiye)

REFERENCES:
- [Background] Davies SJ, Reichardt-Pascal SY, Vaughan D, Russell GI. Differential effect of ischaemia-reperfusion injury on anti-oxidant enzyme activity in the rat kidney. Exp Nephrol. 1995 Nov-Dec;3(6):348-54. PMID 8528679
- [Background] Vafapour M, Nematbakhsh M, Monajemi R, Mazaheri S, Talebi A, Talebi N, Shirdavani S. Effect of Gamma-aminobutyric acid on kidney injury induced by renal ischemia-reperfusion in male and female rats: Gender-related difference. Adv Biomed Res. 2015 Jul 27;4:158. doi: 10.4103/2277-9175.161585. eCollection 2015. PMID 26380243
- [Background] Talebi N, Nematbakhsh M, Monajemi R, Mazaheri S, Talebi A, Vafapour M. The Protective Effect of gamma-aminobutyric Acid on Kidney Injury Induced by Renal Ischemia-reperfusion in Ovariectomized Estradiol-treated Rats. Int J Prev Med. 2016 Jan 11;7:6. doi: 10.4103/2008-7802.173796. eCollection 2016. PMID 26941907